CLINICAL TRIAL: NCT06025084
Title: The Effect of Egg Shell Nanoparticles Combined With Titanium Dioxide Nanoparticles on The Permeability of Dentinal Tubules After Exposure to Wear Challenges and Their Clinical Efficacy in The Treatment of Dentin Hypersensitivity
Brief Title: The Effect of the Egg Shell Nanoparticles Combined With Titanium Dioxide Nanoparticles
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fadia Ali El-Sayed Shosha
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Dentin Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- first group (A1) (Active Comparator): About 24 patients hypersensitive teeth. So the hypersensitive teeth will be treated with egg shell nanoparticles
  Interventions: Drug: Egg Shell nanoparticles
- second group (A2) (Active Comparator): About 24 patients hypersensitive teeth. treated with the combination therapy of eggshell and TiO2.
  Interventions: Drug: Egg Shell nanoparticles

INTERVENTIONS:
Drug: Egg Shell nanoparticles — Evaluate the effects of egg shell nanoparticles combined with Titanium dioxide nanoparticles in the treatment of dentin hypersensitivity at different time intervals.
  Other Names: Titanium dioxide nanoparticles

SUMMARY:
Dentin hypersensitivity is one of the most commonly occurring clinical dental conditions which is characterized by short and sharp pain which arises from exposed dentin in response to external stimuli, which typically are thermal, evaporative, tactile, osmotic or chemical.

Hypersensitive dentin is mostly found in buccal tooth areas, in which enamel is missing because of abrasion, attrition, or erosion. The most generally accepted theory regarding the mechanism of dentin hypersensitivity is the hydrodynamic theory. It proposes that a pain-provoking stimulus increases the flow of the dentinal tubular fluid and consequently, stimulates the nerves around the odontoblasts, leading to dentin hypersensitivity.

DETAILED DESCRIPTION:
Dentin desensitizing products, containing agents such as fluoride, strontium salts, oxalate, glutaraldehyde and bioactive glass, are employed to treat dentin hypersensitivity.

Based on the hydrodynamic theory, there are two main strategies for the treatment of dentin hypersensitivity as: (1) occluding the dentinal tubules to reduce the fluid flow, and (2) decreasing the excitability of the intradental nerve.

Although these products and agents were reported to be effective, short durability and poor effectiveness were often exhibited. The therapeutic effects of these desensitizing products were short lived on account of daily tooth brushing or drinking of acidic beverages and the occlusion effects were sometimes incomplete. Owing to these drawbacks, the use of nanomaterials as dentin occluding material has been predicted to be the future of treating DH.

Amorphous Calcium Phosphate (ACP) has the potential to remineralize the structure of tooth. ACP is a soluble calcium phosphate compound that discharges calcium and phosphate ions to change to apatite and remineralize the tooth structure when it comes in contact with saliva. Forming on the enamel and within the dental tubules, ACP provides a reservoir of phosphate and calcium ions in the saliva Casein phospho-peptide (CPP) is a milk-derived protein that joins to the tooth's biofilm and is applied to stabilize ACP. In recent years, remineralization products used CPP as a vehicle to deliver and preserve a super saturation state of ACP near the surface of tooth. A previous study showed that the application of (CPP-ACP) containing agents as GC tooth mousse and MI paste plus can reduce dentin permeability by occluding dentin tubules. It revealed that these materials can be effective for treatment of dentin hypersensitivity.

Recently, there has been a renewed interest in developing materials with a bioactive potential that could block the exposed dentinal tubules and subsequently reduce the fluid flow within the tubules. Eggshells (EBs) have been investigated in recent years for their remineralization capabilities. EB has rich bioavailable calcium content in the form of carbonates and oxides. It contains 94% calcium carbonate, 1% calcium phosphate, 1% magnesium carbonate, and 4% organic matter. In addition, eggshell provides a cost-effective, renewable, and sustainable source of material for EnHAp. A previous study revealed that eggshell powder is predicted to be the future of tooth remineralization and highly effective in occluding dentinal tubules and reducing dentin hypersensitivity.

Titanium dioxide is one of the few materials that classified as bioactive meaning that it enhances bone growth and stable bone bonding with dental implants via precipitation of hydroxyapatite on its surface

ELIGIBILITY:
Inclusion Criteria:

1- For patients;

* Age between 20 and 55 years
* Patients in good systemic health with clinically elicitable dentin hypersensitivity
* Absence of contraindications to the proposed therapies as allergy. 2 - For teeth;
* Absence of local pathologies (e.g., caries and fractures)
* Visual analog scale (VAS) score ≥3

Exclusion Criteria:

* -- For patients;

  * Use of any desensitizing toothpaste for previous 3 or 4 months.
  * Taking analgesics/anti-inflammatory drugs at the time of the study, pregnancy, and smoking.

    2 -For teeth ;
  * Teeth with abrasion and attrition.
  * Carious lesions on the selected or neighboring teeth, defective restorations
  * Any professional desensitizing therapy on the selected teeth during the last 6 months.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Assessment of dentin hypersensitivity | from baseline to 2 months after the treatment day.
  The pain response will be assessed using the numerical Visual Analogue Scale (VAS, range 0-10), with 0 indicating 'no pain' and 10 indicating 'intolerably severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Hussein, Lecturer, Principal Investigator — Al-Azhar Faculty of Dentistary for girls
Locations (1):
- Faculty of Dentistary - Al-Azhar University, Cairo, Egypt